CLINICAL TRIAL: NCT03246594
Title: Oesophageal Probe Evaluation in RF Ablation of Atrial Fibrillation
Acronym: OPERA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heart Center Leipzig - University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Opera-2016
Record Dates: First submitted 2017-08-08; First posted 2017-08-11 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; esophageal probe; thermolesion
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Esophageal Probe (Experimental): Participants in this group will receive ablation for atrial fibrillation with a oesophageal probe placed for temperature monitoring.
  Placement of oesophageal probe for temperature measurement
  Interventions: Device: Placement of oesophageal probe for temperature measurement
- No Esophageal Probe (Experimental): Participants in this group will receive ablation for atrial fibrillation without a oesophageal probe placed for temperature monitoring.
  Intervention: Power limitation of RF generator
  Interventions: Device: Power limitation of RF generator

INTERVENTIONS:
Device: Placement of oesophageal probe for temperature measurement — The oesophagus probe is used to measure the intraluminal temperature inside the oesophagus
  Arms: Esophageal Probe
Device: Power limitation of RF generator — no probe utilized; Limit the RF Generator Output to 25W
  Arms: No Esophageal Probe

SUMMARY:
The Trial will evaluate the influence of oesophageal probes in Radio frequency (RF)-ablation of atrial fibrillation regarding oesophageal ulcers after ablation.

DETAILED DESCRIPTION:
The Trial will evaluate the influence of oesophageal probes in RF-ablation of atrial fibrillation regarding oesophageal complications after ablation.

200 patients will be prospectively randomised into 2 groups. The conventional group will undergo RF-Ablation of atrial fibrillation using an oesophageal probe to measure the temperature during ablation.

In the other group will receive ablation using fixed energy levels (25 Watt) at the posterior left atrial (LA) Wall without an oesophageal probe , All patients will get a gastroscopy for evaluation of oesophageal complications the day after the procedure.

All patients will have a 6 months follow up (FU) in our clinic to be reevaluated for complications (primary endpoint) and rhythm stability. (secondary endpoint)

ELIGIBILITY:
Inclusion Criteria:

* 12 lead ECG with documented atrial fibrillation
* Indication for RF ablation of atrial fibrillation according to the recent guidelines
* Signed informed consent
* Age 18-85 years

Exclusion Criteria:

* Pregnancy or possible pregnancy without negative test within 48h prior to ablation
* Intracardiac thrombus
* Contraindication for oral anticoagulation
* Conditions, that may complicate the positioning of the oesophageal probe

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-07-03 (Actual); Primary Completion 2019-04-25 (Actual); Study Completion 2019-10-24 (Actual)

PRIMARY OUTCOMES:
Oesophageal complications after RF Ablation depending on using an oesophageal probe | Up to 6 months
  Incidence of oesophageal mucosa alterations in gastroscopy

SECONDARY OUTCOMES:
Rhythm stability after RF ablation of atrial fibrillation (AF) | 6 Months
  Percentage of AF/AT recurrences in 7 day holter at 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Heart Center Leipzig, Leipzig, Germany

REFERENCES:
- [Derived] Schoene K, Arya A, Grashoff F, Knopp H, Weber A, Lerche M, Konig S, Hilbert S, Kircher S, Bertagnolli L, Dinov B, Hindricks G, Halm U, Zachaus M, Sommer P. Oesophageal Probe Evaluation in Radiofrequency Ablation of Atrial Fibrillation (OPERA): results from a prospective randomized trial. Europace. 2020 Oct 1;22(10):1487-1494. doi: 10.1093/europace/euaa209. PMID 32820324